CLINICAL TRIAL: NCT05416125
Title: Lisdexamfetamine for the Treatment of Severe Obesity in Children Aged 6 to 12 Years
Brief Title: Vyvanse in Children Aged 6 to 12 Years
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PEDS-2022-30981
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Obesity, Childhood
Keywords: Obesity
MeSH Terms: conditions — Pediatric Obesity; Obesity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lifestyle therapy plus placebo (Placebo Comparator): Individuals randomized to this arm will receive lifestyle therapy plus placebo for 24 weeks.
  Interventions: Behavioral: Lifestyle therapy
- Lifestyle therapy plus lisdexamfetamine (Active Comparator): Individuals randomized to this arm will receive lifestyle therapy plus lisdexamfetamine for 24 weeks.
  Interventions: Drug: Lisdexamfetamine Dimesylate

INTERVENTIONS:
Drug: Lisdexamfetamine Dimesylate — Vyvanse treatment
  Arms: Lifestyle therapy plus lisdexamfetamine
Behavioral: Lifestyle therapy — Lifestyle treatment
  Arms: Lifestyle therapy plus placebo

SUMMARY:
This study will randomize children who have difficulty maintaining a healthy weight to one of two treatment groups: lifestyle therapy plus lisdexamfetamine or lifestyle therapy plus placebo.

DETAILED DESCRIPTION:
This pilot study will enroll up to 40 children aged 6 to 12 years who have severe obesity. Individuals will be randomized to receive lifestyle therapy plus lisdexamfetamine or lifestyle therapy plus placebo. Participants will receive therapy for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 6 to <12 years at study entry
* Severe obesity defined as BMI >/= 1.2 times the 95th percentile at the screening visit
* Prior failed attempt of lifestyle therapy per parent/guardian report
* Written informed consent of parent/legal guardian and written assent of participant

Exclusion Criteria:

* Contraindications to lisdexamfetamine, including current or recent (< 14 days) use of monoamine oxidase inhibitor and known hypersensitivity to amphetamine products
* Family history of sudden death or ventricular arrhythmia in any first or second degree relative with any of the following: sudden or unexplained death including sudden infant death syndrome, cardiomyopathy, heart transplant, familial arrhythmia (such as Wolff-Parkinson-White syndrome, long QT interval, or implantable defibrillator).
* Any history of fainting or seizure from exercise, startle, or fright
* Clinically significant congenital or structural heart disease or arrhythmia
* BMI <1.2 times the 95th percentile at the baseline/randomization visits
* Hypertension defined as systolic blood pressure (SBP) and/or diastolic blood pressure (DBP) >/= 95th percentile (on 3 separate occasions) at the screening OR baseline/randomization visits
* Tachycardia defined heart rate (HR) >/= 120 bpm (on 3 separate occasions) at the screening OR baseline/randomization visits
* Current or recent (< 3 months) use of psychostimulant or sympathomimetic amine
* History of chemical dependency
* Diabetes mellitus (type 1 or 2)
* Current or recent (< 3 months) use of anti-obesity medication(s)
* Previous bariatric surgery
* Recent initiation or change in dose (< 3 months prior) of anti-hypertensive or lipid medication(s)
* Thyroid stimulating hormone (TSH) > 1.5x upper limit of normal (ULN)
* Aspartate transaminase (AST) or alanine transaminase (ALT) > 3x ULN
* Fasting glucose >/= 126 mg/dL
* History of mania, schizophrenia, bipolar disorder, or psychosis
* Unstable depression or anxiety that has required hospitalization in the past 12 months
* Any history of suicide attempt
* Columbia Suicide Severity Rating Scale (C-SSRS) with a score of Moderate or Hiogh at the screening or baseline/randomization visits
* Children's Depressive Inventory 2 (CDE-2_ score >/= 70 (based on parent or child report) at the screening or baseline/randomization visits
* Concomitant use of tricyclic antidepressants, selective serotonin re-uptake inhibitors (SSRIs), serotonin and norepinephrine re-uptake inhibitors (SNRIs), lithium, fentanyl, tramadol, triptans, tryptophan, buspirone and St. John's wort at any time during the study
* Refusal to use adequate contraception (double barrier method or stable hormonal contraception plus single barrier method, tubal ligation, or abstinence) in girls of childbearing potential
* Inability to swallow test capsule (participants will have two opportunities)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Percent change in Body Mass Index | 24 weeks
  The primary outcome is the percent change in body mass index (BMI) from randomization to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Fox, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT05416125/Prot_SAP_000.pdf
  • Informed Consent Form (2025-06-27): https://cdn.clinicaltrials.gov/large-docs/25/NCT05416125/ICF_001.pdf